CLINICAL TRIAL: NCT01514292
Title: PTL-900590 Effectiveness and Safety Study of the Dexcom G4™ Continuous Glucose Monitoring System
Brief Title: Effectiveness and Safety Study of the Dexcom G4™ Continuous Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTL-900590
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Real Time Continuous Glucose Monitoring System (Experimental): 7 day use of real time continuous glucose monitoring system
  Interventions: Device: Continuous Glucose Monitoring of glucose levels (Dexcom)

INTERVENTIONS:
Device: Continuous Glucose Monitoring of glucose levels (Dexcom) — Manipulation of glucose levels during multiple clinic days. Achieved through diet, exercise and insulin regimen defined in protocol.Evaluation of CGM performance characteristics in reference to a laboratory standard.
  Other Names: CGM System; G4 CGM System; Dexcom G4 CGM System

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of the Dexcom G4 System when used as an adjuvant to blood glucose testing over a 7-day period in people >18 years-old with diabetes mellitus.

The primary objective is to characterize the System performance with respect to laboratory reference venous sample measurements. The device performance will be primarily evaluated in terms of point and rate accuracy of the G4 System in reference to YSI.

Safety of the G4 System will be characterized by Adverse Device Effects and Serious Adverse Device Effects experienced by study participants.

DETAILED DESCRIPTION:
The primary objective is to characterize the System performance with respect to laboratory reference venous sample measurements. The device performance will be primarily evaluated in terms of point and rate accuracy of the G4 System in reference to YSI. The trend accuracy of the device performance, i.e., continuous glucose error grid analysis, will be evaluated as well as the temporal G4 System accuracy at different glucose rates of changes and different glucose ranges (hypoglycemic, euglycemic, and hyperglycemic ranges). The primary matched paired (Sensor-YSI) measurements will be collected during multiple in-clinic days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Diagnosed with diabetes mellitus;
* Use one of the following for their diabetes management:

  * intensive insulin therapy (IIT) or
  * non-intensive insulin therapy (non-IIT)
* Intensive-insulin using (IIT) subjects only - During each in-clinic session, willing to have their blood glucose levels manipulated into high and low glucose levels. Subjects not on IIT will only be observed during each in-clinic session.
* For subjects that exercise routinely (at least 3 times per week), willing to exercise on each in-clinic session, if asked;
* Willing to take a minimum of 7 fingersticks per day during home use days;
* Willing to refrain from the use of acetaminophen during sensor wear period and the day prior to sensor insertion;

Exclusion Criteria:

* Have extensive skin changes/diseases that preclude wearing the required number of devices on normal skin (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis) at the proposed wear sites;
* Have a known allergy to medical-grade adhesives;
* Are pregnant as demonstrated by a positive pregnancy test within 72 hours of sensor insertion,
* Are on dialysis;
* Have a hematocrit that is less than 36% or greater than 55% at screening visit;
* Currently participating in another investigational study protocol (if a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study);
* Have a history of cardiovascular disease (including, but not limited to ischemic heart disease, peripheral vascular disease, cardiomyopathy, cerebrovascular disease, congenital heart disease, or significant arrhythmias), epilepsy, severe migraines in the past 6 months, adrenal disease, syncope, significant hypoglycemia unawareness, or a history of severe hypoglycemia (requiring emergency medical intervention) within the last 6 months;
* Have any chronic infectious disease or intercurrent illness that would interfere with their participation in the study or pose an excessive risk to study staff handling venous or capillary blood samples (e.g. HIV/AIDS, Hepatitis B or C);
* Have a MRI scan, CT scan, or diathermy scheduled during the week of the study. If any of these procedures are required urgently during the study, subjects will notify the study staff, end their CGM session, and remove their sensor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Price, MD, Study Director — DexCom, Inc.
Locations (4):
- United States (4):
  - Profil Institute for Clinical Research, Chula Vista, California
  - AMCR Institute, Inc., Escondido, California
  - Diablo Clinical Research, Walnut Creek, California
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho

RESULTS

PARTICIPANT FLOW:
Groups:
- CGM Device: Dexcom CGM Device Wearing for up to 7 days
Period: Overall Study
Arm/Group | CGM Device
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Type 1 Diabetes and Type 2 Diabetes with Insulin treatment.
Groups:
- Real Time Continuous Glucose Monitoring System: Real Time Continuous Glucose Monitoring(CGM) System Wearing for up to 7 days.
Arm/Group | Real Time Continuous Glucose Monitoring System
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 68
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: CGM Relative Differences to Laboratory Reference
Description: The outcome measure is measured as the relative differences (%) of the CGM glucose value in reference to a laboratory reference, yellow spring instrument( YSI) glucose measurements.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: Percentage of difference
Groups:
- Real Time Continous Glucose Monitoring System: Real Time Continous Glucose Monitoring System Wearing for up to 7 days
Arm/Group | Real Time Continous Glucose Monitoring System
Number analyzed (Participants) | 72
Percentage of difference | 13 (6)
Statistical Analysis 1: Comparison: Real Time Continous Glucose Monitoring System; Hence, the hypothesis is established as: Ho: pi < 71.5% Ha: pi >71.5% Thus, the objective is to conclude that the proportion of G4 Sensor-YSI points in the present study meeting the 20 mg/dL/20% criterion is no worse than the existing FDA-approved SEVEN PLUS System. The null hypothesis will be rejected if pi observed in this study is greater than 71.5%, the G4 System performance is no worse than the historical performance of the existing FDA approved CGM system will be concluded; Test type: Superiority or Other; p = 0.0001, Fisher Exact

ADVERSE EVENTS:
Time Frame: 7 day use of continuous glucose monitoring system
Arm/Group | CGM Device
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No